CLINICAL TRIAL: NCT06849102
Title: Effects of NeuroReAlign Therapy on Balance and Gait in Stroke Survivors: a Randomized Controlled Trial
Brief Title: NeuroReAlign Therapy for Balance and Gait Rehabilitation in Stroke Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Middle East University (Other)
Responsible Party: Principal Investigator, Anas Radi Hassan Alashram, Assistant Professor, Middle East University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADA/1099
Record Dates: First submitted 2025-02-20; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Physiotherapy (Active Comparator): Patients in this group will receive conventional physiotherapy interventions, including treadmill training, balance training, strengthening and stretching lower limb muscles, for 45 minutes per session, 3 times weekly, for 4 weeks.
  Interventions: Other: conventional physiotherapy interventions
- NeuroReAlign Therapy (Experimental): Patients in this group will receive NeuroReAlign Therapy, including motor training (e.g., treadmill training, balance training), multimodal sensory stimulation (e.g., proprioceptive and visual), cognitive training (e.g., traditional cognitive exercise), and motivation, for 45 minutes per session, 3 times weekly, for 4 weeks.
  Interventions: Other: NeuroReAlign Therapy

INTERVENTIONS:
Other: NeuroReAlign Therapy — Patients in this group will receive NeuroReAlign Therapy, including motor training (e.g., treadmill training, balance training), multimodal sensory stimulation (e.g., proprioceptive and visual), cognitive training (e.g., traditional cognitive exercise), and motivation, for 45 minutes per session, 3 times weekly, for 4 weeks.
  Arms: NeuroReAlign Therapy
Other: conventional physiotherapy interventions — Patients in this group will receive conventional physiotherapy interventions, including treadmill training, balance training, strengthening and stretching lower limb muscles, for 45 minutes per session, 3 times weekly, for 4 weeks.
  Arms: Conventional Physiotherapy

SUMMARY:
The goal of this randomized controlled trial is to investigate the effects of NeuroReAlign Therapy on balance and gait in stroke survivors in the chronic stage (>6 months). The study will include male and female participants aged 18-70 years.

The main questions it aims to answer are:

Does NeuroReAlign Therapy improve balance in stroke survivors compared to conventional physiotherapy? Does NeuroReAlign Therapy enhance gait performance more effectively than conventional physiotherapy? Researchers will compare NeuroReAlign Therapy to conventional physiotherapy to determine its effects on balance and gait.

Participants will:

Undergo NeuroReAlign Therapy or conventional physiotherapy for 4 weeks. Have their balance assessed using the Berg Balance Scale (BBS), Activities-Specific Balance Confidence Scale (ABC Scale), and Fear of Falling Questionnaire (FoFQ).

Have their gait evaluated using the Dynamic Gait Index (DGI), Rivermead Mobility Index (RMI), Timed Up and Go (TUG), 6-Minute Walk Test (6MWT), and 10-Meter Walk Test (10MWT).

Complete outcome assessments at baseline and after the intervention (week 4).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic or hemorrhagic stroke
* Have a stroke more than 6 months
* Age between 18 and 70

Exclusion Criteria:

* Patients with severe cognitive impairments
* Patients cannot walk independently

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Dynamic Gait Index (DGI) | At baseline (week 0) and after the intervention (week 4)
  The Dynamic Gait Index (DGI) is a clinical tool designed to assess an individual's ability to adapt gait to varying task demands, particularly in populations with neurological conditions such as stroke, Parkinson's disease, and vestibular disorders. It consists of eight walking-related tasks, including changes in gait speed, head movements, obstacle navigation, and stair climbing, each scored on a 4-point scale (0-3), with a maximum total score of 24. Lower scores indicate greater impairment and a higher risk of falls, with a cutoff score of ≤19 suggesting increased fall risk. The DGI is widely used in rehabilitation settings to evaluate functional mobility, guide treatment planning, and monitor progress in individuals with balance and gait deficits.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | At baseline (week 0) and post-intervention (week 4)
  The Berg Balance Scale (BBS) is a widely used clinical assessment tool designed to evaluate balance in individuals, particularly in older adults or those with neurological conditions such as stroke. It consists of 14 tasks that assess a range of balance activities, including sitting, standing, reaching, turning, and stepping. Each task is scored on a scale from 0 to 4, with a maximum total score of 56. A higher score indicates better balance, while lower scores suggest a greater risk of falling. The BBS is a reliable and valid tool for both clinical assessments and monitoring balance over time, making it a key measure in rehabilitation settings for individuals with balance impairments.
Activities-Specific Balance Confidence Scale (ABC Scale) | At baseline (week 0) and post-intervention (week 4)
  The Activities-Specific Balance Confidence Scale (ABC Scale) is a self-reported measure used to assess an individual's confidence in maintaining balance while performing various daily activities. The scale consists of 16 items, each asking the participant to rate their confidence (on a percentage scale from 0% to 100%) in performing specific tasks, such as walking, climbing stairs, or moving around the house, without losing balance or becoming unsteady. A higher score reflects greater confidence in balance, while lower scores indicate fear of falling or instability. The ABC Scale is widely used in clinical settings to evaluate balance confidence, identify fall risk, and track changes over time, especially in populations with balance and mobility impairments, such as those recovering from stroke or other neurological conditions.
Fear of Falling Questionnaire (FoFQ) | At baseline (week 0) and post-intervention (week 4)
  The Fear of Falling Questionnaire (FoFQ) is a clinical tool used to assess an individual's fear of falling, which is often associated with decreased mobility, balance issues, and increased fall risk. It consists of several questions that explore the level of concern a person has about falling in various situations, such as walking in different environments or performing daily activities. The questionnaire typically uses a Likert scale to rate the intensity of fear, with higher scores indicating greater fear of falling. The FoFQ helps identify individuals at risk of avoiding activities due to fear of falling, which can lead to reduced physical function and further decline in mobility. It is widely used in rehabilitation and geriatric care to assess fear of falling, guide interventions, and monitor progress in patients with balance disorders or neurological conditions.
Rivermead Mobility Index (RMI) | At baseline (week 0) and post-intervention (week 4)
  The Rivermead Mobility Index (RMI) is a clinical assessment tool used to measure mobility in individuals with neurological conditions, particularly those recovering from stroke or other brain injuries. It consists of 15 items that evaluate a range of mobility tasks, such as sitting, standing, walking, and transferring between different positions. Each task is scored on a scale from 0 to 15, with higher scores indicating greater mobility. The RMI is designed to assess both basic functional movements and more complex mobility tasks, making it suitable for tracking changes in functional ability over time. It is a reliable and valid measure widely used in rehabilitation settings to evaluate and monitor recovery progress, guide treatment plans, and predict outcomes in individuals with mobility impairments.
Timed Up and Go (TUG) | At baseline (week 0) and post-intervention (week 4)
  The Timed Up and Go (TUG) test is a simple and widely used clinical assessment tool to evaluate mobility, balance, and fall risk in individuals, particularly those with neurological conditions or the elderly. The test involves timing how long it takes a person to rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down again. The total time taken to complete the task is recorded, with longer times indicating poorer mobility and a higher risk of falling. The TUG is a quick, efficient, and reliable test that can be used to assess functional mobility in various clinical and rehabilitation settings, offering valuable insights into an individual's ability to perform basic mobility tasks independently.
10-Meter Walk Test (10MWT) | At baseline (week 0) and post-intervention (week 4)
  The 10-Meter Walk Test (10MWT) is a widely used clinical measure to assess walking speed and gait function in individuals, particularly in those with neurological conditions or mobility impairments. The test involves timing how long it takes a person to walk a distance of 10 meters at their usual pace, and the walking speed is calculated by dividing the time taken by the distance. The 10MWT is a reliable indicator of mobility and can be used to assess walking performance, identify walking abnormalities, and evaluate improvements over time, making it especially useful in rehabilitation and clinical settings. Faster times generally indicate better functional mobility, while slower times may suggest gait difficulties or higher fall risk.
6-Minute Walk Test (6MWT) | At baseline (week 0) and post-intervention (week 4)
  The 6-Minute Walk Test (6MWT) is a simple, reliable, and widely used outcome measure that assesses a person's walking endurance and functional capacity. During the test, participants are instructed to walk as far as possible over a 6-minute period on a flat, hard surface, typically a 30-meter or 50-foot corridor. The distance covered within the allotted time is recorded as the primary outcome. The 6MWT evaluates not only gait speed but also the individual's cardiovascular and muscular endurance, making it an important tool for assessing the overall functional mobility of individuals, particularly those with neurological or musculoskeletal disorders, such as stroke. It is commonly used to assess the effects of interventions like rehabilitation or exercise training on walking endurance, and can also be used to monitor progress or decline over time.